CLINICAL TRIAL: NCT02606331
Title: Evaluation the Efficacy of Flapless Corticotomy Accomplished by Either Hard-laser or Piezosurgey in Accelerating Upper Canine Retraction and Evaluation of the Dento-alveolar Changes and the Levels of Acceptance and Discomfort.
Brief Title: Efficacy of Minimally Invasive Surgical Technique in Accelerating Orthodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-03-2015
Record Dates: First submitted 2015-11-11; First posted 2015-11-17 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Malocclusion, Angle Class II
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Piezosurgery; Lasers, Solid-State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Piezosurgery (Experimental): In one half of the dental arch, piezosurgery will be performed for canine retraction, whereas in the other half ordinary canine retraction procedure will be followed.
  Interventions: Procedure: Piezosurgery
- ER:YAG Laser (Experimental): In one half of the dental arch, ER:YAG laser irradiation will be performed for canine retraction, whereas in the other half ordinary canine retraction procedure will be followed.
  Interventions: Radiation: ER:YAG laser

INTERVENTIONS:
Procedure: Piezosurgery — Corticotomy cuts will be performed by this technique.
  Arms: Piezosurgery
Radiation: ER:YAG laser — Corticotomy cuts will be performed by this technique.
  Arms: ER:YAG Laser

SUMMARY:
Thirty six patients needs therapeutic extraction of the maxillary first premolars with subsequent retraction of the maxillary canines will be divided randomly into two groups : piezocision group and the ER:yttrium aluminum garnet (YAG) laser group. In each group, piezocision or hard laser-assisted flapless corticotomy will randomly assigned to one side of the maxillary arch at the first premolar region, and the other side served as the control. Canine retraction will be initiated after completion of the leveling and alignment phase via closed nickel-titanium coil springs applying 150 g of force per side, soldered trans-palatal arch will be used as an anchor unit.

Pre- and post distalization dental casts will be evaluated to study rate of canine distalization, canine rotation and anchorage loss over a follow-up period until a Class I canine relationship is achieved. The levels of pain and discomfort will be self-reported using a questionnaire with visual analog scales administered at four assessment times during the first month after the minimally invasive procedure.

DETAILED DESCRIPTION:
One main issue in orthodontics is the prolonged treatment time, leading patients, especially adults, to avoid treatment or seek alternative options such as implants or veneers with less than optimal results.

Therefore, the search for methods that decrease the treatment duration is a main challenge in orthodontic research. Decreased duration of therapy seems to be related not only to better patient compliance, but also to reduced treatment -related root resorption , better periodontal health and lower risk of caries and white spots. Adjunct to the proper selection of brackets, wires, biomechanic systems, force levels, and anchorage systems, an array of novel techniques has been introduced to accelerate orthodontic tooth movement. These techniques can be briefly categorized as surgical and non-surgical. However The surgical approach is the most clinically used and most tested with known predictions and stable results. The invasiveness of surgical procedures, requiring full mucoperiosteal flaps, might have been a drawback for their widespread acceptance among orthodontists and patients. Therefore, more conservative flapless corticotomy techniques have recently been proposed. Although various techniques of flapless corticotomy have been reported to be successful in practice, scientific evidence for their effectiveness so far has been limited to case series and a handful of clinical trials, generally with small groups. Therefore further controlled prospective studies are needed to study the effectiveness of flapless corticotomy in accelerating orthodontic tooth movement .

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy patients , Male and female , Age range: 15-27 years.
* Class II Division 1 malocclusion :

  * Mild / moderate skeletal Class II (sagittal discrepancy angle ≤7)
  * Overjet ≤10
  * Normal or excessive facial height (Clinically and then cephalometrically assessed using these three angles : mandibular/cranial base angle, maxillary/mandibular plane angle and facial axis angle)
  * Mild to moderate crowding ≤ 4
* Permanent occlusion.
* Existence of all the upper teeth (except third molars).
* Good oral and periodontal health:

  * Probing depth < 4 mm
  * No radiographic evidence of bone loss .
  * Gingival index ≤ 1
  * Plaque index ≤ 1

Exclusion Criteria:

* Medical problems that affect tooth movement (corticosteroid, nonsteroidal antiinflammatory drugs (NSAIDs), …)
* patients have anti indication for oral surgery ( medical - social - psycho)
* Presence of primary teeth in the maxillary arch
* Missing permanent maxillary teeth (except third molars).
* Poor oral hygiene or Current periodontal disease:

  * Probing depth ≥ 4 mm
  * radiographic evidence of bone loss
  * Gingival index > 1
  * Plaque index > 1
* Patient had previous orthodontic treatment

Ages: 14 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Rate of canine retraction | This will be measured immediately at the end of the tooth movement, i.e. when the retracted canine reaches its final position which takes up to 12 weeks
  The distance traveled by mm is divided by the time required in weeks.

SECONDARY OUTCOMES:
Rate of molar anchorage loss | This will be measured immediately at the end of the tooth movement, i.e. when the retracted canine reaches its final position which may take up to 12 weeks
  The amount of mesial movement of the first molar in millimeters (mm) is divided by the time required to retract the upper canines (in weeks).
Change in canine rotation | This will be measured at the following assessment times: T1: baseline, T2: after 4 weeks of canine retraction, T3: after 8 weeks of canine retraction, T4: when the canine reaches its final position up to 12 weeks
  This measurement will be performed on plaster models taken at the aforementioned assessment times.
Change in the levels of pain and discomfort | These levels will be assessed at: one day following the intervention, one week, two weeks, and four weeks following the intervention.
  Assessment will be performed using questionnaires via visual analog scales.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Alfawal, DDS, Principal Investigator — MSc student at the Orthodontic Department, University of Damascus Dental School; Mohammad Y Hajeer, DDS MSc PhD, Study Chair — Associate Professor of Orthodontics, University of Damascus Dental School
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Rif-dimashq Governorate, Syria

REFERENCES:
- [Background] Aksakalli S, Calik B, Kara B, Ezirganli S. Accelerated tooth movement with piezocision and its periodontal-transversal effects in patients with Class II malocclusion. Angle Orthod. 2016 Jan;86(1):59-65. doi: 10.2319/012215-49.1. Epub 2015 May 19. PMID 25989211
- [Background] Alikhani M, Raptis M, Zoldan B, Sangsuwon C, Lee YB, Alyami B, Corpodian C, Barrera LM, Alansari S, Khoo E, Teixeira C. Effect of micro-osteoperforations on the rate of tooth movement. Am J Orthod Dentofacial Orthop. 2013 Nov;144(5):639-48. doi: 10.1016/j.ajodo.2013.06.017. PMID 24182579
- [Background] Al-Naoum F, Hajeer MY, Al-Jundi A. Does alveolar corticotomy accelerate orthodontic tooth movement when retracting upper canines? A split-mouth design randomized controlled trial. J Oral Maxillofac Surg. 2014 Oct;72(10):1880-9. doi: 10.1016/j.joms.2014.05.003. Epub 2014 May 14. PMID 25128922
- [Background] Aboul-Ela SM, El-Beialy AR, El-Sayed KM, Selim EM, El-Mangoury NH, Mostafa YA. Miniscrew implant-supported maxillary canine retraction with and without corticotomy-facilitated orthodontics. Am J Orthod Dentofacial Orthop. 2011 Feb;139(2):252-9. doi: 10.1016/j.ajodo.2009.04.028. PMID 21300255
- [Background] Hoogeveen EJ, Jansma J, Ren Y. Surgically facilitated orthodontic treatment: a systematic review. Am J Orthod Dentofacial Orthop. 2014 Apr;145(4 Suppl):S51-64. doi: 10.1016/j.ajodo.2013.11.019. PMID 24680025
- [Derived] Alfawal AMH, Hajeer MY, Ajaj MA, Hamadah O, Brad B. Evaluation of piezocision and laser-assisted flapless corticotomy in the acceleration of canine retraction: a randomized controlled trial. Head Face Med. 2018 Feb 17;14(1):4. doi: 10.1186/s13005-018-0161-9. PMID 29454369